CLINICAL TRIAL: NCT05543746
Title: Dynamic Neural Mechanisms of Brexanolone-induced Antidepressant Effects in Postpartum Depression: a Feasibility Study
Brief Title: Dynamic Neural Mechanisms of Brexanolone-induced Antidepressant Effects in Postpartum Depression
Acronym: BRX-PPD
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Baszucki Brain Research Fund (Other); Sage Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-2224
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Brexanolone — Enrolled subjects will receive a 60-hour infusion of Brexanolone (BRX) according to FDA approved protocol for administration. A programmable peristaltic infusion pump will be used to ensure accurate delivery.
  Other Names: Zulresso

SUMMARY:
This is a feasibility study of performing repeated EEG recordings and assessment of affective states during open-label administration of BRX to women with postpartum depression. Study phases will include screening, enrollment, intervention, and follow-up. Subjects will be screened for study eligibility criteria through clinical assessments and self-report. Enrolled subjects will be admitted to the UNC Women's Hospital, where five serial EEG recordings will be obtained, along with frequent assessments of affective state, before, during, and after a 60-hour IV infusion of BRX. Follow-up procedures will include assessments of PPD and affective symptoms, as well as an exit interview with the study team. If feasibility outcomes are achieved, exploratory EEG analyses will be performed with AMICA (adaptive mixture independent component analysis), community detection, and microstate assessment. Exploratory analyses of data collected by facial expression detection software (iMotions Affectiva) are also planned.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Documented proof of full COVID-19 vaccination
* Ambulatory, female, aged 18-45
* ≤ 8 months postpartum
* Agrees to adhere to the study requirements.
* Onset of depression in 3rd trimester or within 4 weeks of delivery
* Meets DSM-V criteria for major depressive disorder with peripartum onset.
* 17-item HAM-D total score ≥20 at screening
* Stopped breastfeeding or agrees to temporarily stop for 7 days including 4 days of hospitalization and 3 days after
* No new psychotropic drugs during screening and active treatment of study
* Stable use of any current psychotropic drugs for at least 28 days prior to enrollment, with stable dosage for at least 14 days prior to enrollment
* Must be on documented contraceptive.
* Must have a caregiver or family member with them to help care for the subject's child(ren) during the infusion and to be in the room with the subject if the child(ren) are present during the infusion

Exclusion Criteria:

* Positive pregnancy test at screening or day 1
* Pregnancy that resulted in a stillbirth, termination, or child that was placed for adoption.
* Renal impairment or failure, hepatic impairment or failure, or anemia
* Untreated or inadequately treated hypothyroidism or hyperthyroidism
* Known allergy to progesterone or allopregnanolone.
* Suicide attempt at this episode
* Medical history of schizophrenia, and/or schizoaffective disorder
* Current psychotic symptoms including delusions, hallucinations, or formal thought disorder.
* Concurrent substance abuse
* Exposure to another investigational medication or device within 30 days
* Has previously participated in any study employing brexanolone or SAGE-217.
* Subject is investigative site personnel, sponsor personnel, or an immediate member of their family.
* Has received electroconvulsive therapy during current episode.
* History of seizure disorder
* On anticonvulsant agents
* On benzodiazepines

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with moderate to severe PPD, medically eligible to receive FDA-approved BRX infusion, recruited from current inpatient and outpatient population in the Women's Mood Disorders Clinic at UNC and through local advertisements. Subjects recruited from outpatient setting will be individuals for whom BRX is the chosen recommended course of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Girdler, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Brexanolone: Based on an FDA-approved regimen, the 60-hour infusion was administered as follows: 30 mcg/kg/hour (Hour 0 to 4), then 60 mcg/kg/hour (Hour 4 to 24), then 90 mcg/kg/hour (Hour 24 to 52), followed by 60 mcg/kg/hour (Hour 52 to 56), and 30 mcg/kg/hour (Hour 56 to 60).
Period: Overall Study
Arm/Group | Brexanolone
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Successfully Analyzed EEG Recordings
Description: Feasibility of EEG recordings. Each participant was scheduled to have 5 EEG recordings.
Time Frame: 4 days
Measure: Number; unit: EEG recordings
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
EEG recordings | 49

2. Primary Outcome: Number of Subjects Completing the Entire Study Protocol Through the Follow-up Phase
Description: Feasibility of study completion
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
Participants | 10

3. Primary Outcome: Number of Subjects Withdrawn From Protocol Due to Adverse Events or Participation Burden
Description: Feasibility of subject burden
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of follow-up period (up to Day 30)
Arm/Group | Brexanolone
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brexanolone (N=10)
Dizziness (Nervous system disorders) | 4 (4)
Fatigue (General disorders) | 3 (3)
Dry mouth (General disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (4)
Infusion site bruising (General disorders) | 2 (2)
Infusion site pain (General disorders) | 2 (2)
Flushing (Vascular disorders) | 4 (4)
Difficulty concentrating (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT05543746/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT05543746/ICF_001.pdf